CLINICAL TRIAL: NCT03005249
Title: Neural Stem Cells Therapy for Cerebral Palsy: a Prospective, Randomized, Parallel-controlled Trial
Brief Title: Neural Stem Cells Therapy for Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Liu Jing, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCKY2016-60
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neural stem cells therapy group (Experimental): The patients will be assigned to neural stem cells therapy group for cerebral palsy.
  Interventions: Procedure: neural stem cells therapy group
- the control group (Experimental): The patients will be assigned to the control group for cerebral palsy.
  Interventions: Other: the control group

INTERVENTIONS:
Procedure: neural stem cells therapy group — The patients will be assigned to neural stem cells therapy group for cerebral palsy.
  Arms: neural stem cells therapy group
Other: the control group — The patients will be assigned to the control group for cerebral palsy.
  Arms: the control group

SUMMARY:
To evaluate the safety and efficacy of neural stem cells (NSCs) therapy for cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is the most severe lifelong disability disease in childhood. In China, an epidemiological investigation of cerebral palsy in 2004 has reported that 2.74‰ (about 6.50-9.75 million) of children suffered from cerebral palsy. The costs of medical expenses, living allowance and nursing care can go up to RMB 20000-50000 yuan per year for each child with cerebral palsy and thus China will expend RMB 120-300 billion yuan per year for children with cerebral palsy. With full liberalization of two-child policy, there is an increasing number of second babies born to women who are 35 years or older. Thus, the incidence of cerebral palsy tends to increase. There is currently no cure for cerebral palsy, resulting in a heavy burden for families and on society. Recent clinical trials performed in countries outside China have demonstrated that stem cell therapy is likely the most effective method to treat cerebral palsy. Fifteen trials regarding stem cell therapy for cerebral palsy have been registered with ClinicalTrials.gov. In China, there have been no standardized registered trials regarding stem cell therapy for cerebral palsy, which greatly restricts its clinical application. In October 2016, the National Health and Family Planning Commission and the Food and Drug Administration of China jointly announced the premier stem cell clinical research institutions, making performing standardized trials regarding stem cell therapy for cerebral palsy in China possible.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with ischemic/hypoxic cerebral palsy (mainly including neonate with asphyxia and premature infants);
* Clinical manifestation of spastic tetraplegia;
* With moderate to severe cerebral palsy, The Gross Motor Function; Classification System (GMFCS) levels IV-V;
* Age 1-5 years, of either sex;
* Provision of signed informed consent by one of his/her parents or legal guardians prior to commencement of this study;

Exclusion Criteria:

* Systemic diseases that possibly influence treatment or patient's compliance;
* Potentially life-threatening diseases involving various organ systems;
* Brain deformity;
* Abnormal behaviors or mood disorder;
* Allergies from blood products;
* Suffering from infectious disease;
* Subjected to craniocerebral operations prior to screening.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
GMFM-88 score | changes of month 1, month 3, month 6, month 9 and month 12 after therapy
  To evaluate change in gross motor function in children with cerebral palsy.

SECONDARY OUTCOMES:
Fine Motor Function Measure (FMFM) score | changes of month 1, month 3, month 6, month 9 and month 12 after therapy
  To evaluate change in fine motor function in children with cerebral palsy.
Modified Ashworth Scale score | changes of month 1, month 3, month 6, month 9 and month 12 after therapy
  To measure resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Ph.D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lv Z, Li Y, Wang Y, Cong F, Li X, Cui W, Han C, Wei Y, Hong X, Liu Y, Ma L, Jiao Y, Zhang C, Li H, Jin M, Wang L, Ni S, Liu J. Safety and efficacy outcomes after intranasal administration of neural stem cells in cerebral palsy: a randomized phase 1/2 controlled trial. Stem Cell Res Ther. 2023 Feb 9;14(1):23. doi: 10.1186/s13287-022-03234-y. PMID 36759901